CLINICAL TRIAL: NCT02346682
Title: Neurochemical,Metabonomics and Neuroimaging Characterization of TCM Diagnostic Subtypes of Major Depression Disorder
Brief Title: Neurochemical, Metabonomics and Neuroimaging Characterization of TCM Diagnostic Subtypes of Major Depression Disorder
Acronym: NMNTDM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Provincial Tongde Hospital (Other)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lan-ying Liu, associate chief physician, Zhejiang Provincial Tongde Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: zjsltdyy2014009; 8140151401 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2014-12-18; First posted 2015-01-27 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2015-04

CONDITIONS: Severe Major Depression Disorder
Keywords: major depression disorder; biochemistry; TCM diagnosis; Neurological; metabonomics; neuroimaging
MeSH Terms: conditions — Neurologic Manifestations | interventions — Venlafaxine Hydrochloride; Clonazepam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- LDQS group (Active Comparator): Liver Depression and Qi Stagnation (LDQS)group,Liver Depression and Qi Stagnation Syndrome should include at least the following 5 symptoms and signs: emotional depression or sadness, pessimism, short breath, sigh, dysphoria，thin coating，stringy pulse Drugs use generic name :Venlafaxine; Dosage form:capsule Dosage, frequency and duration:Venlafaxine dose was initiated at 75 mg/day and escalated to an optimal dose (150-225 mg/day in most cases) within 2 week, depending upon individual patient response, but the maximum dose could not exceed 300 mg/day during the next 4 weeks.
  The biomarkers of neurobiochemistry, metabonomics and neuroimaging would be tested at the baseline and after 6-week venlafaxine administration.
  Interventions: Drug: venlafaxine
- DBHS group (Active Comparator): Deficiency of Both Heart and Spleen (DBHS) group,Deficiency of Both Heart and Spleen Syndrome should include at least following 6 symptoms and signs: emotional depression, thinking torpidity, tiredness, forgetfulness, insomnia, loose stool, sweating, pale tongue body, thin tongue coating, and thin and deep pulse Drugs use generic name :Venlafaxine; Dosage form:capsule Dosage, frequency and duration:Venlafaxine dose was initiated at 75 mg/day and escalated to an optimal dose (150-225 mg/day in most cases) within 2 week, depending upon individual patient response, but the maximum dose could not exceed 300 mg/day during the next 4 weeks.
  The biomarkers of neurobiochemistry, metabonomics and neuroimaging would be tested at the baseline and after 6-week .
  Interventions: Drug: venlafaxine
- the normal controls group (No Intervention): The normal controls group including the healthy volunteer None drug The biomarkers of neurobiochemistry, metabonomics and neuroimaging would be tested at the baseline .

INTERVENTIONS:
Drug: venlafaxine — Venlafaxine dose was initiated at 75 mg/day and escalated to an optimal dose (150-225 mg/day in most cases) within 2 week, depending upon individual patient response, but the maximum dose could not exceed 300 mg/day during the next 4 weeks. Patients were prescribed a combination of venlafaxine and Benzodiazepines for sleep disturbance.
  Other Names: clonazepam
  Arms: DBHS group; LDQS group

SUMMARY:
There is heterogeneity in patients with depression. Many scholars propose that individualization of antidepressant achieves better outcomes. However, the scientific theoretical basis of individualized treatment is still quite weak. Different clinical subtypes of depression and their possible biomarkers are critically needed to provide the individualization with theoretical base. Diagnostic types of major depression disorder (MDD) based on the Theory of Traditional Chinese Medicine (TCM) and possible differentiations in neurobiochemistry, metabonomics and neuroimaging could be one of ways to explore the biomarkers and support the theory of the individualized treatment.

The hypothesized results will be of help to clarify the biological basis of MDD with LDQS and with DBHS, to provide the TCM with further scientific evidence, to explore the pathogenesis of depression, to improve the objective diagnosis of depression, and to promote targeted interventions by Western medicine, TCM or both.

DETAILED DESCRIPTION:
The objectives of this study is to explore if there are any differences in neurobiochemistry, metabonomics and neuroimaging (1) at the baseline, between the subjects who are the normal controls (C Group) and who both meet diagnostic criteria of the Diagnostic and Statistical Manual of 5th edition (DSM-V) on MDD and TCM criteria of 'pattern of Liver Depression and Qi Stagnation (LDQS)' or'pattern of Deficiency of Both Heart and Spleen (DBHS)' (T Group); (2) at the baseline, between the MDD subjects of LDQS and DBHS; (3) after 6-week venlafaxine administration, between the MDD subjects of LDQS and DBHS. 50 subjects in T Group and 25 in C Group are recruited in the study and the main laboratory tests include High Performance Liquid Chromatography(HPLC), Gas Chromatography-Mass Spectrum(GCMS) and neuroimaging DTI technology.

ELIGIBILITY:
Inclusion Criteria:

1. Had a diagnosis of major depressive disorder according to DSM-V and TCM criteria of 'pattern of Liver Depression and Qi Stagnation (LDQS)' or'pattern of Deficiency of Both Heart and Spleen (DBHS)
2. The severity of the symptoms is moderate or severe, confirmed by a 35 or greater of Hamilton Rating Scale for Depression(HAMD) score
3. Absence of brain and/or severe physical diseases
4. 18-65years old

Exclusion Criteria:

1. In pregnancy，brain and other severe medical conditions
2. Psychoactive substance abuse
3. Had a diagnosis of bipolar disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Brain neuroimaging | 2 years
  Diffusion Tensor Imaging(DTI) is used to detect changes in FA maps of brain white matter fiber in major depressive patients

SECONDARY OUTCOMES:
Biochemical tests | 2 years
  Gas Chromatography-Mass Spectrum is used to test blood and urine samples for:
  lactic acid, alanine, 3 - hydroxy butyric acid, valine, carbamide, glycerinum, phosphoric acid, isoleucine, glycine, succinic acid, threonine, malic acid, glutamic acid, citric acid, stearic acid, GABA, methionine, cysteine, lysine, tryptophan, leucine, methionine and tyrosine.

OTHER OUTCOMES:
Neurochemical tests | 2 years
  High Performance Liquid Chromatography (HPLC) is used to detect blood samples for:
  5-HT, NE, DA, 5-HTAA, and HVA.

CONTACTS AND LOCATIONS:
Overall Officials: Lan-ying Liu, Master, Study Director — Zhejiang Provincial Tongde Hospital
Locations (1):
- Tongde hospital of zhejiang province, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Liu LY, Xu XP, Luo LY, Zhu CQ, Li YP, Wang PR, Zhang YY, Yang CY, Hou HT, Cao YL, Wang G, Hui ES, Zhang ZJ. Brain connectomic associations with traditional Chinese medicine diagnostic classification of major depressive disorder: a diffusion tensor imaging study. Chin Med. 2019 Apr 11;14:15. doi: 10.1186/s13020-019-0239-8. eCollection 2019. PMID 31044001
- [Derived] Liu LY, Zhang HJ, Luo LY, Pu JB, Liang WQ, Zhu CQ, Li YP, Wang PR, Zhang YY, Yang CY, Zhang ZJ. Blood and urinary metabolomic evidence validating traditional Chinese medicine diagnostic classification of major depressive disorder. Chin Med. 2018 Oct 25;13:53. doi: 10.1186/s13020-018-0211-z. eCollection 2018. PMID 30386416